CLINICAL TRIAL: NCT01983527
Title: A Prospective Randomized 3-arm Trial Comparing Intra-articular Corticosteroid Injection vs Arthrographic Distention vs Arthrographic Distention Plus Intra-articular Corticosteroid Injection in the Treatment of Adhesive Capsulitis
Brief Title: Corticosteroids and / or Arthrographic Distention in the Treatment of Adhesive Capsulitis
Acronym: CADAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imelda Hospital, Bonheiden (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Symons Rolf, Symons Rolf, MD, Imelda Hospital, Bonheiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CADAC
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
Keywords: Arthrographic distention; Hydrodilatation; Intra-articular corticosteroid injection
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arthrographic distention + intra-articular corticosteroid (Experimental): Arthrographic distention of the glenohumeral joint with injection of 5 ml contrast, 1 ml (40 mg) Depo Medrol(Methylprednisolone Acetate Injectable Suspension), 15 ml local anaesthetic (Prilocaine) and up to 15 ml saline.
  Interventions: Procedure: Arthrographic distention; Drug: Intra-articular corticosteroid Depo Medrol
- Arthrographic distention (Active Comparator): Arthrographic distention of the glenohumeral joint with injection of 5 ml contrast, 15 ml local anaesthetic (Prilocaine) and up to 15 ml saline.
  Interventions: Procedure: Arthrographic distention
- Intra-articular corticosteroid (Active Comparator): Arthrographic pseudodistention of the glenohumeral joint with injection of 5 ml contrast and 1 ml (40 mg) Depo Medrol(Methylprednisolone Acetate Injectable Suspension).
  Interventions: Drug: Intra-articular corticosteroid Depo Medrol

INTERVENTIONS:
Procedure: Arthrographic distention — Arthrographic distention of the glenohumeral joint with injection of 5 ml contrast, 15 ml local anaesthetic (Prilocaine) and up to 15 ml saline.
  Other Names: Hydrodilatation
  Arms: Arthrographic distention; Arthrographic distention + intra-articular corticosteroid
Drug: Intra-articular corticosteroid Depo Medrol — Intra-articular injection of 1 ml (40 mg) Depo Medrol(Methylprednisolone Acetate Injectable Suspension)
  Arms: Arthrographic distention + intra-articular corticosteroid; Intra-articular corticosteroid

SUMMARY:
Arthrographic distention of the shoulder joint is an increasingly popular treatment option in the management of patients with frozen shoulder. Most have included the intra-articular injection of a corticosteroid as part of the procedure, but it is not known if this is necessary. It is also not known whether arthrographic distention using steroid and saline is better than intra-articular steroid injection alone.

The purpose of this study is to determine whether there is an additional benefit in the combination of arthrographic distention plus intra-articular corticosteroid injection compared to arthrographic distention or intra-articular corticosteroid injection alone.

ELIGIBILITY:
Inclusion Criteria:

* Pain and stiffness in predominantly 1 shoulder for 4 weeks or longer
* Restriction of passive motion of greater than 30° in 2 or more planes of movement (measured to onset of pain with goniometer)

Exclusion Criteria:

* Previous arthrographic distention and/or corticosteroid injection
* Systemic inflammatory joint disease
* Radiological evidence of osteoarthritis of the shoulder or fracture
* Signs of a complete rotator cuff tear
* Contraindications to arthrogram and/or distention
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index(SPADI) | 4 weeks

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | weekly for a period of 3 months plus at follow-up (4 months and 12 months)
Overall pain score | weekly for a period of 3 months, plus at follow-up (4 months and 12 months)
  Universal pain scale
Range of motion | 4 weeks, 4 months and 12 months
  * Total shoulder abduction (in degrees, measured with goniometer)
  * External rotation in neutral position (in degrees, measured with goniometer)
  * Hand behind back (highest reachable anatomical landmark)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Symons, MD, Principal Investigator — Imeldaziekenhuis
Locations (1):
- Imelda Hospital, Bonheiden, Antwerpen, Belgium

REFERENCES:
- [Background] Jacobs LG, Barton MA, Wallace WA, Ferrousis J, Dunn NA, Bossingham DH. Intra-articular distension and steroids in the management of capsulitis of the shoulder. BMJ. 1991 Jun 22;302(6791):1498-501. doi: 10.1136/bmj.302.6791.1498. PMID 1855018
- [Background] Corbeil V, Dussault RG, Leduc BE, Fleury J. [Adhesive capsulitis of the shoulder: a comparative study of arthrography with intra-articular corticotherapy and with or without capsular distension]. Can Assoc Radiol J. 1992 Apr;43(2):127-30. French. PMID 1562888
- [Background] Gam AN, Schydlowsky P, Rossel I, Remvig L, Jensen EM. Treatment of "frozen shoulder" with distension and glucorticoid compared with glucorticoid alone. A randomised controlled trial. Scand J Rheumatol. 1998;27(6):425-30. doi: 10.1080/030097498442244. PMID 9855212
- [Background] Buchbinder R, Green S, Forbes A, Hall S, Lawler G. Arthrographic joint distension with saline and steroid improves function and reduces pain in patients with painful stiff shoulder: results of a randomised, double blind, placebo controlled trial. Ann Rheum Dis. 2004 Mar;63(3):302-9. doi: 10.1136/ard.2002.004655. PMID 14962967
- [Background] Khan AA, Mowla A, Shakoor MA, Rahman MR. Arthrographic distension of the shoulder joint in the management of frozen shoulder. Mymensingh Med J. 2005 Jan;14(1):67-70. PMID 15695959